CLINICAL TRIAL: NCT06892548
Title: A Phase Ib/II, Multi-site, Open-label, Two-part Trial to Evaluate the Efficacy, Safety, Pharmacokinetics, and Recommended Combination Dose of BNT324 With BNT327 in Participants With Advanced Lung Cancer
Brief Title: A Clinical Study to Investigate the Efficacy and Safety of an Investigational Combination Therapy With BNT324 and BNT327 in Patients With Advanced Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: DualityBio Inc. (Industry); Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BNT324-01; 2024-520238-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-19; First posted 2025-03-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced Lung Cancer
Keywords: Small cell lung cancer (SCLC); Non-small cell lung cancer (NSCLC); Programmed death-ligand 1 (PD-L1); Vascular endothelial growth factor (VEGF); Bispecific antibody; BNT324 (DB-1311); BNT327; Combination with chemotherapy; Combination with other investigational agents; Immunotherapy; Treatment-naïve
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1 - BNT324 + BNT327 combination therapy (Experimental): Escalating combination dose levels of BNT324 and BNT327 to define RP2D and RP2D-1 for NSCLC and SCLC.
  Interventions: Biological: BNT324; Biological: BNT327
- Part 2 - Cohort 1: RP2D of BNT324 + BNT327 and RP2D-1 of BNT324 + BNT327 (Experimental): In subpopulation 1 of NSCLC actionable oncogenic alteration (AGA) negative, first-line (1L)
  Interventions: Biological: BNT324; Biological: BNT327
- Part 2 - Cohort 2: RP2D of BNT324 + BNT327 and RP2D-1 of BNT324 + BNT327 (Experimental): In SCLC, second-line plus (2L+)
  Interventions: Biological: BNT324; Biological: BNT327
- Part 2 - Cohort 3: RP2D of BNT324 + BNT327 (Experimental): In subpopulation 1 of NSCLC AGA negative, 2L+
  Interventions: Biological: BNT324; Biological: BNT327
- Part 2 - Cohort 4: RP2D of BNT324 + BNT327 (Experimental): In subpopulation 2 of NSCLC AGA negative, 1L
  Interventions: Biological: BNT324; Biological: BNT327
- Part 2 - Cohort 5: RP2D of BNT324 + BNT327 (Experimental): In subpopulation 2 of NSCLC AGA negative, 2L+
  Interventions: Biological: BNT324; Biological: BNT327
- Part 2 - Cohort 6: RP2D of BNT324 + BNT327 (Experimental): In NSCLC AGA positive
  Interventions: Biological: BNT324; Biological: BNT327
- Part 2 - Cohort 7: RP2D of BNT324 + BNT327 (Experimental): In SCLC, 1L
  Interventions: Biological: BNT324; Biological: BNT327

INTERVENTIONS:
Biological: BNT324 — Intravenous infusion
  Other Names: DB-1311
Biological: BNT327 — Intravenous infusion

SUMMARY:
This study aims to investigate the combination of BNT324, a B7-H3 antibody-drug conjugate (ADC) with BNT327, a programmed death-ligand 1 (PD-L1) and vascular endothelial growth factor (VEGF) bispecific antibody, in participants with advanced/metastatic or relapsed/progressive small cell lung cancer (SCLC) and non small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a two-part study designed to evaluate and establish two safe combination dose levels (recommended Phase 2 dose [RP2D] and a lower/another combination dose level [RP2D-1]) of BNT324 with BNT327 (Part 1), to determine the optimal combination dose (dose optimization [DO]) in NSCLC and SCLC lead indication cohorts at the RP2D and RP2D-1, to evaluate the preliminary efficacy in selected lung cancer cohorts at the highest combination dose level (in a signal seeking Part 2), and to confirm the clinical efficacy of BNT324 in combination with BNT327 at the optimal dose level in participants with advanced lung cancer in expansion cohorts (proof-of-concept [POC] cohorts).

The study consists of a screening period, a treatment period, a safety follow-up period, and a long-term survival follow-up period.

In Part 1 participants with histologically or cytologically confirmed relapsed or progressive lung cancer (both SCLC and NSCLC are eligible) will receive BNT324 in combination with BNT327 using a dose escalation design.

In Part 2 of the study, BNT324 will be studied in combination with BNT327 at the RP2D compared to RP2D-1 in participants with advanced metastatic treatment-naïve NSCLC (DO Cohort 1) and relapsed/progressive SCLC after failure of cytotoxic chemotherapy with or without immuno-oncology (IO) (DO Cohort 2). The totality of the available data (e.g., safety, efficacy, pharmacokinetics etc.) will be reviewed to select the optimal dose. After the optimal dose is selected, additional participants in each cohort may be enrolled in the selected optimal dose.

In the signal seeking cohorts (Cohort 3-7), participants will receive BNT324 in combination with BNT327 at the RP2D from Part 1.

A predefined number of participants in Part 2 Cohort 1 and Cohort 2 will be randomized to one of the two dose levels (RP2D and RP2D-1) selected from Part 1 in a 1:1 ratio. Additional participants in Part 2 Cohort 1 and Cohort 2 may be enrolled in the selected optimal dose to further assess the efficacy and safety profile.

No randomization is planned for any other cohort in Part 2 or Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at the time of giving informed consent.
* Histological or cytological confirmed unresectable advanced/metastatic lung cancer. Histological classification may be based on tumor samples prior to metastatic disease. Participants with mixed histology must be classified based on the main component. Participants with NSCLC are eligible with any or no PD-L1 expression. Participants with AGA-positive disease must have received targeted therapy prior to enrollment in this study.

  * Part 1: Participants with NSCLC and SCLC
  * Part 2 Cohort 1: Participants with NSCLC (subpopulation 1) AGA negative, 1L
  * Part 2 Cohort 2: Participants with SCLC, 2L+
  * Part 2 Cohort 3: Participants with NSCLC (subpopulation 1) AGA negative, 2L+
  * Part 2 Cohort 4: Participants with NSCLC (subpopulation 2) AGA negative, 1L
  * Part 2 Cohort 5: Participants with NSCLC (subpopulation 2) AGA negative, 2L+
  * Part 2 Cohort 6: Participants with NSCLC AGA positive
  * Part 2 Cohort 7: Participants with SCLC, 1L
* Have measurable disease defined by RECIST version 1.1.
* Have an Eastern Cooperative Oncology Group performance status of 0 or 1.
* Have a life expectancy of ≥12 weeks.

Exclusion Criteria:

* Prior treatment with B7-H3 targeted therapy.
* Prior treatment with ADC with topoisomerase inhibitor (e.g., datopotamab deruxtecan, trastuzumab deruxtecan). Note: This exclusion applies to participants in the first-line/treatment-naïve cohorts in the advanced/metastatic setting. Prior treatment with ADC with topoisomerase inhibitor payload is only allowed for participants in the second-line plus cohorts in the advanced/metastatic setting.
* Is a candidate to locoregional treatment (including surgical resection, stereotactic radiotherapy or tumor ablation) with potential to induce complete or near complete response and prolonged tumor control (sometimes described as "radical" intent), per investigator's assessment.
* Has a history of significant hematologic toxicity to prior lines of therapy, as assessed by investigator, e.g., Grade 4 febrile neutropenia or recurrent/persistent Grade 3 to 4 neutropenia.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply to all or some participants depending on the cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Occurrence of dose limiting toxicities (DLTs) by dose level | During the DLT evaluation period, i.e., the time of initiation of the first dose of investigational medicinal product (IMP) up to 21 days]
Part 1 - Occurrence of Treatment-emergent adverse events (TEAEs), serious TEAEs, treatment-related TEAEs, and treatment-related serious TEAEs by dose level | From the time of the first dose of IMP to 90 days after the last IMP dose or until new anticancer therapy is started, whichever occurs first
Part 1 - Occurrence of dose interruption, reduction, and treatment discontinuations due to TEAEs by dose level | From the time of the first dose of IMP to 90 days after the last dose of IMP or until new anticancer therapy is started, whichever occurs first
Part 2 cohorts 1 and 2 - Occurrence of TEAEs, serious TEAEs, treatment-related TEAEs, and treatment-related serious TEAEs by cohort and treatment arm | From the time of the first dose of IMP to 90 days after the last IMP dose or until new anticancer therapy is started, whichever occurs first
Part 2 cohorts 1 and 2 - Occurrence of dose interruption, reduction, and treatment discontinuation due to TEAEs by cohort and treatment arm | From the time of the first dose of IMP to 90 days after the last IMP dose or until new anticancer therapy is started, whichever occurs first
Part 2 cohorts 1 and 2 - Objective response rate (ORR) by cohort and treatment arm | From the time of initiation of the first dose of IMP to end of study, i.e., up to 87 months
  ORR defined as the proportion of participants in whom a confirmed complete response (CR) or partial response (PR) is observed as best overall response (per response evaluation criteria in solid tumors [RECIST] version 1.1 based on the investigator's assessment).
Part 2 cohorts 3-7 - ORR by cohort | From the time of initiation of the first dose of IMP to end of study, i.e., up to 87 months
  ORR, defined as the proportion of participants in whom a confirmed CR or PR is observed as best overall response (per RECIST version 1.1 based on the investigator's assessment).

SECONDARY OUTCOMES:
Part 1 - ORR by dose level | From the time of initiation of the first dose of IMP to end of study, i.e., up to 87 months
  ORR, defined as the proportion of participants in whom a confirmed CR or PR is observed as best overall response (per RECIST version 1.1 based on the investigator's assessment).
Part 1 - Disease control rate (DCR) by dose level | From the time of initiation of the first dose of IMP to end of study, i.e., up to 87 months
  DCR, defined as the proportion of participants with confirmed CR, PR, or stable disease (SD) as best overall response (per RECIST version 1.1 based on the investigator's assessment).
Part 2 all cohorts - (PFS) by cohort and treatment arm | From the time of initiation of the first dose of IMP to end of study, i.e., up to 87 months
  PFS defined as the time from first dose of IMP to the first objective tumor progression (PD) or death from any cause, whichever occurs first, per RECIST version 1.1 based on the investigator's assessment.
Part 2 all cohorts - Duration of response (DOR) by cohort and treatment arm | From the time of initiation of the first dose of IMP to end of study, i.e., up to 87 months
  DOR, defined as the time from first objective response (CR or PR) to first occurrence of objective tumor progression (PD) or death from any cause, whichever occurs first (per RECIST version 1.1 based on the investigator's assessment).
Part 2 all cohorts - Overall survival (OS) by cohort and treatment arm | From the time of initiation of the first dose of IMP to end of study, i.e., up to 87 months
  OS, defined as the time from first dose of IMP to death from any cause.
Part 2 all cohorts - DCR by cohort and treatment arm | From the time of initiation of the first dose of IMP to end of study, i.e., up to 87 months
  DCR, defined as the proportion of participants with confirmed CR, PR, or SD as best overall response (per RECIST version 1.1 based on the investigator's assessment).
Part 2 all cohorts - Time to response (TTR) by cohort and treatment arm | From the time of initiation of the first dose of IMP to end of study, i.e., up to 87 months
  TTR, defined as the time from first dose of IMP to first objective response (CR or PR per RECIST version 1.1 based on the investigator's assessment).
Part 2 cohorts 3-7 - Occurrence of TEAEs, serious TEAEs, treatment-related TEAEs, and treatment-related serious TEAEs by cohort and treatment arm | From the time of the first dose of IMPs to 90 days after the last IMP dose or until new anticancer therapy is started, whichever occurs first
Part 2 cohorts 3-7 - Occurrence of dose interruption, reduction, and treatment discontinuation due to TEAEs by cohort and treatment arm | From the time of the first dose of IMP to 90 days after the last IMP dose or until new anticancer therapy is started, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (45):
- United States (12):
  - Precision NextGen Oncology and Research Center, Beverly Hills, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA - David Geffen School of Medicine, Santa Monica, California
  - University of Iowa Hospitals & Clinics PARENT, Iowa City, Iowa
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York
  - Icahn School of Medicine at Mount Sinai PRIME, New York, New York
  - Cleveland Clinic Taussig Cancer Institute Case Comprehensive Cancer Center, Cleveland, Ohio
  - Texas Oncology - DFW, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - Northeast, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Australia (5):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Bendigo Hospital, Bendigo, Victoria
  - Barwon Health, Geelong, Victoria
  - Sunshine Hospital, Saint Albans, Victoria
  - St John of God Subiaco Hospital, Subiaco, Western Australia
- China (16):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing GoBroad Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi Zhuang
  - The First Affiliated Hospital of Xinxiang Medical University, Weihui, Henan
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Linyi Cancer Hospital, Shandong, Linyi
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai GoBroad Cancer Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (5):
  - Adana City Hospital, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Dr. Abdurrahman Yurtaslan Oncology Teaching and Research Hospital, Ankara
  - Ankara City Hospital, Ankara
  - Yeditepe University Medical School Hospital, Istanbul
- United Kingdom (3):
  - Bristol Haematology and Oncology Centre, Bristol
  - St. James's University Hospital, Leeds
  - University College London Hospital, London

IPD SHARING:
Plan to Share IPD: No